CLINICAL TRIAL: NCT05348850
Title: Correlation Between Contractile Properties of Quadriceps Muscle and Functional Performance in Runners With Patellofemoral Pain Syndrome
Brief Title: Quadriceps Muscle Contractile Properties and Functional Performance
Status: Completed | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Menan Aliy Eldeen Mohamed Elmahdy, Principal Investigator, Cairo University
Other Study IDs: P.T.REC/012/003382
Record Dates: First submitted 2022-04-13; First posted 2022-04-27 (Actual); Last update posted 2023-01-17 (Actual); Status verified 2023-01

CONDITIONS: Patellofemoral Pain Syndrome
Keywords: Runners
MeSH Terms: conditions — Patellofemoral Pain Syndrome

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Study Group: Athletes with patellofemoral pain syndrome will be selected Muscle contractile properties and functional performance will be assessed for athletes with patellofemoral pain syndrome .
  Data will be collected from all athletes regarding age, gender, training intensity running experience and previous injuries.
  By the end of the assessment it will be detected if muscle contractile properties of vastus medialis and vastus lateralis is a determinant factor that influence functional performance in runners with patellofemoral pain syndrome.
  Interventions: Device: Tensiomayography (TMG)

INTERVENTIONS:
Device: Tensiomayography (TMG) — Quadriceps muscle contractile properties will be assessed using tensiomayography

SUMMARY:
The aim of this study is to investigate the association between tensiomyography parameters (from rectus femoris, vastus lateralis and vastus medialis) and functional abilities in runners with patellofemoral pain syndrome.

DETAILED DESCRIPTION:
Running is one of the most widespread activities during which overuse injuries of the lower extremity occur. Long-distance running is very popular among participants of recreational sports . In 2008, about 11.5% of the population in the United States ran and, of this group, 3.4% ran on average two times a week or more. In Europe, it is estimated that 36% of the population aged 15-65 years are recreational runners.

Most running-related injuries occur in the lower extremities. The most common anatomical site of running injuries is the knee.

Risk factors for running injuries have been well investigated , However, because of the heterogeneity of the studies (e.g., definition of injury, recreational or elite runners, and short- or long-distance runners), no clear overview is available regarding the most important risk factors for running injuries. Increased training volume per week in male runners, and a history of previous injuries for runners, are known significant risk factors for running injuries.

The various purported risk factors for running injuries are commonly divided into intrinsic and extrinsic risk factors. Intrinsic risk factors include mostly anatomic and other variables that are innate to the individual, such as gender, age, height, weight, personality type (e.g., aggressive, passive), and anatomic factors such as femoral anteversion, genu varus or valgus, pes planus or cavus, bone density, muscular flexibility, and leg-length discrepancies. Extrinsic risk factors include training variables such as mileage, hill running, pace, interval training, equipment (shoes, shoe inserts), and training surfaces.

Patellofemoral pain syndrome is the most common overuse injury of the lower extremity, and is particularly prevalent in those who are physically active. For example, approximately 2.5 million runners will be diagnosed with PFPS in a given year. PFPS also is a significant problem in the military as it has been reported that 37% of recruits develop PFPS while in basic combat training. Females are reported to be at greater risks for PFPS than their male counterparts. Alarmingly, 70% to 90% of individuals with PFPS have recurrent or chronic pain, In addition, the result of a recent study suggest that having PFPS as a younger individual may predispose one to develop patellofemoral osteoarthritis later in life.

One of the most common risk factors of patellofemoral pain syndrome is the imbalance of the quadriceps musculature and maltracking of the patella are 2 potential factors that may lead to PFP.

The nature of PFP is multifactorial, and many risk factors have been associated with this condition. This come in agreement with several authors who reported that patellofemoral pain syndrome is one of the most common injuries in runners.

ELIGIBILITY:
Inclusion Criteria:

* The athletes age range between 18-30 years old will participate in this study.
* Both males and females will participate in this study.
* All athletes will be selected from long-distance runners.
* All athletes have an average running period (6 days per week and 5 hours per day).

Exclusion Criteria:

* Athletes with foot deformities such as hallux valgus, foot supination, pes planus, and pes cavus,
* Athletes with biomechanical abnormalities and complications affecting walking ability and performance.
* History of lower limbs or back surgery or injury.
* Structural or functional leg length discrepancy.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: 30 Distance runners selected from Egyptian clubs will participate in the study.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2022-04-20 (Actual); Primary Completion 2022-09-20 (Actual); Study Completion 2023-01-01 (Actual)

PRIMARY OUTCOMES:
Contractile properties of Quadriceps muscle for 30 runners with patellofemoral pain syndrome | measured at the baseline as it is a cross sectional study
  Will be assessed using Tensiomayography
Anteromedial lunge Functional Performance Test designed for 30 runners with patellofemoral pain syndrome | measured at the baseline as it is a cross sectional study
  Anteromedial lunge test will be performed by each athlete for 3 trails with a 3 min recovery period between .
Step-down Functional Performance Test designed for 30 runners with patellofemoral pain syndrome | measured at the baseline as it is a cross sectional study
  Step-down test will be performed by each athlete for 3 trails with a 3 min recovery
Balance and reach Functional Performance Test designed for 30 runners with patellofemoral pain syndrome | measured at the baseline as it is a cross sectional study
  Balance and reach test will be performed by each athlete for 3 trails with a 3 min recovery

CONTACTS AND LOCATIONS:
Overall Officials: kahled ayad, Prof, Study Chair — Professor of Orthopaedic Physical Therapy, Deraya University and Cairo University, Egypt
Locations (1):
- Haven Health care, El-Sheikh Zayed City, Egypt

IPD SHARING:
Plan to Share IPD: Undecided